CLINICAL TRIAL: NCT04710238
Title: Assessment of Gonadal Functions in Hemodialysis Male Patients on Regular Hemodialysis :A Cross-Sectional Study.
Brief Title: Assessment of Gonadal Functions in Uremic Male Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Setohy Hussein Ali, Resident physician ,internal medicine departement , nephrology unite, Assiut University
Other Study IDs: uremic hypogonadism
Record Dates: First submitted 2020-09-27; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: ESRD
Keywords: uremic hypogonadism; free testosterone level; serum prolactin
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Study the prevalence of sexual dysfunction in male patients on hemodialysis aged 18-60 years (sexually active male) .
2. Study the effect of hemodialysis on the male patients sexual functions by measurement of serum prolactin and free testosterone levels.

DETAILED DESCRIPTION:
: Gonadal dysfunction is a frequent finding in men with ESRD on chronic hemodialysis ,erectile dysfunction is one of the most common manifestation of sexual dysfuncion whitch has been reported to be as high as 70 -80 %of hemodialysis patients .

Testosterone deficiency and insufficiency are frequent findings in hemodialysis male patients that were found to be 66% and 24% respectively The Probleme is multifactorial , the most important factor is due to testesterone deficiency. total and free testosterone levels are typically reduced , that is usually accompanied by elevation of serum Gonadotropins concentrations due to hypothalamic -pituitary-gonadal -axis disturbance(uremic hypogonadism) .

Alterations in the pulsatile release of GnRH, which leads to a hypogondal state due to uremia, which occurs due to inadequate nutrient intake, stress, and systemic illness . Excess LH secretion is thought to result from the diminished release of testosterone from the Leydig cells, because testosterone normally provides a feedback inhibition of LH release. The metabolic clearance rate of LH is reduced due to reduction of kidney clearance ,Follicle stimulating hormone (FSH) secretion is also increased in men with chronic kidney failure.

Elevated plasma prolactin levels are commonly found in dialyzed men, it is thought to be due to increased its production , extreme hyperprolactinemia has been associated with infertility, loss of libido, low circulating testosterone levels, So,due to testosterone deficiency and hyperprolactinemia in ESRD as one of most important factors and exclusion of other factors , men on chronic hemodialysis shows different degrees of subfertility or infertility due to Erectile dysfunction , testicular damage and impaired spermatogenesis.

ELIGIBILITY:
* Inclusion Criteria

  1. Male patients.
  2. ESRD on chronic hemodialysis with GFR lower than 15ml/min /1.73 m2
  3. Age (18_60)years old
* Exclusion Criteria:

  1-Diabetic patients . 3-hypertesive patients . 3-Patients with primary infertility before the event of ESRD and Starting dialysis.

  4-Manifest hypothyroidism . 5-Patient with other causes that may lead to subfertility as varicocele . 6-patients with previous exposure to head and genital trauma , surgery or irradiation .

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male patients aged 18-60 (sexualy active males )
Study Population: male patients that were diagnosed to be ESRD on hemodialysis , newly diagnosed and patients on chronic hemodialysis for years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Study the prevalence of sexual dysfunction in male patients on hemodialysis . | base line
  Knowning the degree of sexual dysfunctions prevalence in male patients on hemodialysis and evaluation of the associated factors of gonadal dysfunction in male patients on hemodialysis .

REFERENCES:
- [Background] Palmer BF, Clegg DJ. Gonadal dysfunction in chronic kidney disease. Rev Endocr Metab Disord. 2017 Mar;18(1):117-130. doi: 10.1007/s11154-016-9385-9. PMID 27586847
- [Background] Antonucci M, Palermo G, Recupero SM, Bientinesi R, Presicce F, Foschi N, Bassi P, Gulino G. Male sexual dysfunction in patients with chronic end-stage renal insufficiency and in renal transplant recipients. Arch Ital Urol Androl. 2016 Jan 14;87(4):299-305. doi: 10.4081/aiua.2015.4.299. PMID 26766802
- [Background] Foulks CJ, Cushner HM. Sexual dysfunction in the male dialysis patient: pathogenesis, evaluation, and therapy. Am J Kidney Dis. 1986 Oct;8(4):211-22. doi: 10.1016/s0272-6386(86)80029-4. PMID 3532769
- [Result] Fiuk JV, Tadros NN. Erectile dysfunction in renal failure and transplant patients. Transl Androl Urol. 2019 Apr;8(2):155-163. doi: 10.21037/tau.2018.09.04. PMID 31080776